CLINICAL TRIAL: NCT06484413
Title: Repetitive Transcranial Magnetic Stimulation for Depression
Brief Title: rTMS for Depression
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS16-0437
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rTMS Group: received rTMS

SUMMARY:
This is a longitudinal observational study, where we will track outcomes in patients undergoing 5 weeks of FDA approved right DLPFC rTMS treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 to 80 years of age
2. DSM V diagnosis of a major depressive episode Subjects must have an initial score of at least 20 on the HAMD at screen
3. rTMS is clinically indicated
4. Patient is competent to provide informed consent

Exclusion Criteria:

1. Lifetime DSM-V diagnosis of schizophrenia, schizoaffective disorder, psychotic depression or any other psychotic disorder as defined in the DSM-V
2. Current (within the last year) diagnosis of anxiety disorder, obsessive- compulsive disorder, or eating disorder that precedes the onset of the current episode of depression and is the primary diagnosis
3. Current diagnosis of delirium, dementia, or amnestic amnesiac disorder
4. Diagnosis of mental retardation
5. Baseline Mini Mental State Exam (MMSE) score < 21 or a total score falling two standard deviations below the age- and education-adjusted mean, whichever is less
6. Any active general medical condition or CNS disease which can affect cognition or response to treatment
7. Current (within the past three months) diagnosis of active substance dependence, or active substance abuse within the past week as indicated by self-report.
8. ECT or rTMS within three months
9. Pregnancy as indicated by self-report
10. MRI contraindications
11. Implanted electronic device or metal implant in the head and neck region (DBS, cochlear implant, etc)
12. Change in the dose of psychotropic medications within the past week

Inclusion Criteria for healthy volunteers:

1. Male or female between age 18 and 80
2. Patient is competent to provide informed consent

Exclusion Criteria for healthy volunteers:

1. Lifetime history of major chronic mental illness, such as schizophrenia, major depression, or bipolar disorder
2. Lifetime history of psychiatric hospitalization because of any mental illness Mental illness, other than depression, that needed psychological or pharmacological treatment in the past
3. Any neurodevelopmental or neurodegenerative disease, or stroke or positive findings on past head CT or brain MRI
4. Pregnancy
5. Hamilton Rating Scale for Depression (HRSD-17) is more than 7
6. MRI contraindications

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female patients with a major depressive episode who are referred for an acute course of rTMS as part of their standard of care will be recruited for the study. Recruitment will occur at The Zucker Hillside Hospital at Northwell Health.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
MADRS | 5 weeks
  Montgomery-Asberg Depression Rating Scale

IPD SHARING:
Plan to Share IPD: Undecided